CLINICAL TRIAL: NCT03078595
Title: Is Gingival Bleeding a Symptom of Patients With Type 2 and 3 Von Willebrand Disease? A Case-Control Study
Brief Title: Gingival Bleeding and Von Willebrand Disease Typ 2 and 3
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Peter Eickholz, Head of Periodontology, Goethe University
Other Study IDs: 143/15
Record Dates: First submitted 2017-03-01; First posted 2017-03-13 (Actual); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Gingival Bleeding; Von Willebrand Diseases
Keywords: periodontal disease; plaque-induced gingivitis; bleeding on probing; von willebrand disease; gingival bleeding
MeSH Terms: conditions — Gingival Hemorrhage; von Willebrand Diseases; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- von Willebrand disease type 2 and 3: Examinations (haematologically and periodontally) of von Willebrand disease patients with type 2 and 3 and healthy controls to evaluate whether type 2 and 3 VWD determines an increased susceptibility to gingival bleeding in response to the oral biofilm
- controls: For each case (VWD) a respective haematologically healthy control is recruited from the gingivitis and periodontitis patients of the Department of Periodontology, Centre for Dentistry and Oral Medicine (Carolinum), Johann Wolfgang Goethe-University Frankfurt/Main. Each control is matched to one of the respective cases for sex, age (±5 years), self-reported smoking status (current smoker/non-smoker), number of remaining teeth (±2 teeth), and periodontal diagnosis (gingivitis, chronic or aggressive periodontitis).

SUMMARY:
Von Willebrand disease (VWD) is the most common inherent bleeding disorder resulting in prolonged bleeding time. Gingival bleeding is a frequently reported symptom of VWD. However, gingival bleeding is also known as a leading symptom of plaque-induced gingivitis and untreated periodontal disease. Gingival bleeding in VWD patients may be triggered by gingival inflammation and not a genuine symptom. Thus, this study evaluates whether type 2 and 3 VWD determines an increased susceptibility to gingival bleeding in response to the oral biofilm.

DETAILED DESCRIPTION:
Patients

All patients with type 2 and 3 VWD consecutively consulting the Haemophilia Centre, Medical Clinic III/Institute for Transfusion medicine, Hospital of the Johann Wolfgang Goethe-University Frankfurt/Main are asked to participate in this study as cases. They are asked for bleeding and subjective symptoms indicating periodontal disease.

The study complies with the rules of the Declaration of Helsinki and was approved by the Institutional Review Board for Human Studies of the Medical Faculty of the Goethe-University Frankfurt/Main (Application# 143/15). All participating individuals are informed on risks and benefits as well as the procedures of the study and give written informed consent.

Controls

For each case (VWD) a respective hematologically healthy control is recruited from the gingivitis and periodontitis patients of the Department of Periodontology, Centre for Dentistry and Oral Medicine (Carolinum), Johann Wolfgang Goethe-University Frankfurt/Main. Each control is matched to one of the respective cases for sex, age (±5 years), self-reported smoking status (current smoker/non-smoker), number of remaining teeth (±2 teeth), and periodontal diagnosis (gingivitis, chronic or aggressive periodontitis).

All participants are asked about current and past cigarette smoking habits. Patients who report smoking or have quit smoking for less than five years are classified as smokers. Additionally the amount of carbon monoxide (CO) in exhaled air is measured using a device (Bedfont Smokerlyzer; Bedfont Scientific Ltd, Rochester, Great Britain).

Hematologic examinations

20 ml of blood are sampled from an arm vein. The following data are assessed at the Haemophilia Centre for clinical routine during VWD patient care and due to study design in the controls:

* von Willebrand parameters (VWF antigen [VWF:Ag], Ristocetin cofactor [VWF:RCo], coagulation factor VIII [FVIII:C])
* Current medication if any VWF:Ag and VWF:RCo were measured turbidimetrically using a device (BCS, Siemens, Marburg, Germany). FVIII:C was assessed with specific agents on a coagulation analyser (ACL-300®, Instrumentation Laboratory, Kirchheim, Germany).

Periodontal examinations

The following clinical parameters are assessed at 6 sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual):

* modified Gingival Bleeding Index (GBI)
* modified Plaque Control Record (PCR)
* PPD and recession to the nearest 0.2 mm using an electronic probe (Florida Probe, Version 3.2, Gainesville, USA). Recession is assessed from the cemento-enamel junction (CEJ) to the gingival margin. At sites where the CEJ was destroyed by restorations the restoration margin (RM) is used as reference. At sites where the CEJ or RM is located apically from the gingival margin the value for recession is negative
* Bleeding on probing (BOP) recorded as positive when bleeding occurs within 30 seconds from probing. For each patient a BOP index is calculated providing the amount of sites with positive BOP in % per patient.

Attachment loss (PAL-V) is calculated as sum of PPD and recession.

All individuals are classified into the following diagnoses:

* plaque-induced gingivitis (PPD < 3.6 mm; PAL-V ≤ 2 mm),
* generalized mild, localized moderate chronic periodontitis (PPD ≥ 3.6 mm; vertical probing attachment level [PAL-V] 3 to 4 mm ≤ 30% of sites; 1 to 2 mm > 30% of sites),
* generalized mild, localized severe chronic periodontitis (PPD ≥ 3.6 mm; PAL-V ≥ 5 mm ≤ 30% of sites; 1 to 2 mm > 30% of sites)
* generalised moderate chronic periodontitis (PPD ≥ 3.6 mm; PAL-V 3 to 4 mm > 30%)
* generalised moderate localised severe chronic periodontitis (PPD ≥ 3.6 mm; PAL-V 3 to 4 mm > 30%; ≥ 5 mm ≤ 30%)

In all individuals hematological and periodontal examinations are obtained within 24 hours. After dental and periodontal examination all patients receive oral hygiene instructions and professional tooth cleaning. In cases of untreated periodontal disease periodontal treatment is offered. VWD are asked to report any bleeding complications after periodontal probing and professional tooth cleaning.

Statistical analysis

The individual patient is used as statistical unit. All analyses are performed on patient level. GBI is defined as the main outcome variable and BOP as secondary outcome variable. All other parameters are control variables. Up to now there are no studies comparing GBI or BOP between VWD type 2 and 3 cases and hematologically healthy controls and there are no standard deviations of mean GBI and BOP for cases and controls. To detect a clinically relevant inter-group difference of 4% GBI or BOP with a type 1 error alpha < 0.05 and a test power of 80% with a standard deviation of group means of 5.5% a sample size of at least 31 individuals is required per group. Thus, it was decided to recruit 31 VWD cases and respectively matched 31 controls.

For all individuals, cigarette pack years are calculated. Group frequencies (VWD, control) are expressed for sex, current smoking. Group means and standard deviations are calculated for GBI, BOP, age, number of remaining teeth, pack years, CO, PCR, VWF:Ag, VWF:RCO, FVIII:C. Further, for each individual the following variables are calculated to describe the periodontal status:

* Mean±standard deviation of PPD and PAL-V
* Percentage of PPD < 4 mm, 4 to 6.8 mm, ≥ 7 mm
* Sum of all PPD, i.e. the sum of the PPD measured at all sites within a patient
* Sum of all PPD with BOP, ), i.e. the sum of the PPD measured at all sites exhibiting BOP within a patient
* Periodontal inflamed surface area (PISA). For each patient PPD were entered into an Excel sheet that can be downloaded freely (http://www.parsprototo.info/pisa.html).

From these group means and standard deviations are calculated. Comparisons between groups for dichotomous parameters are made by χ² or Fisher's exact test and for all other parameters by Mann-Whitney-U test. A post-hoc analysis is performed to estimate the test power that would be required to find a clinically relevant inter-group difference (δ) of 5% for GBI and BOP index with a type 1 error (α) of 0.05 for the actual sample size.

Using stepwise linear backward multiple regression analysis, factors shall be identified that influence GBI and BOP. The following independent variables are entered into the model for GBI: group (VWD/control), sex, age, number of remaining teeth, PCR, CO, pack years, PISA. The following independent variables are entered into the model for BOP: group (VWD/control), sex, age, number of remaining teeth, PCR, CO, pack years, PISA. Due to the fact that mean PPD is mathematically coupled to sum of PPD, sum of PPD with BOP, and PISA these 4 variables are not entered into the regression model at the same time. PISA provides the best representation of the subgingival inflamed area. Thus, PISA is chosen for the final model. The following parameters are described by dummy variables: group (control = 0, VWD = 1), sex (male = 0, female = 1), smoking status (never and former smoker = 0, current smoker = 1). All factors with p < 0.1 are kept in the models. For statistical analysis a PC program is used (SystatTM for Windows Version 12, Systat Inc., Evanston, USA).

ELIGIBILITY:
Inclusion Criteria von Willebrand Patients:

* 18 - 80 years old
* no other bleeding disorder except 2 and 3 von Willebrand disease

Inclusion Criteria healthy controls:

* no bleeding disorder
* no anticoagulative medication

Exclusion Criteria von Willebrand Patients:

- requirement of systemic antibiotics for measures that may cause transitory bacteraemia

Exclusion Criteria healthy controls:

- bleeding disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases with type 2 and 3 VWD consecutively consulting the Haemophilia Centre, Medical Clinic III/Institute for Transfusion medicine, Hospital of the Johann Wolfgang Goethe-University Frankfurt/Main are asked to participate in this study as cases. For each case (VWD) a respective haematologically healthy matched control is recruited from the gingivitis and periodontitis patients of the Department of Periodontology, Centre for Dentistry and Oral Medicine (Carolinum), Johann Wolfgang Goethe-University Frankfurt/Main.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Eickholz, Prof., Study Chair — Dept. of Perio, Center for Dent. and Oral Med., JWG-University Frankfurt
Locations (2):
- Germany (2):
  - Center for Dentistry and Oral Medicine (Carolinum), Johann Wolfgang Goethe-University, Frankfurt am Main, Hesse
  - Dept. of Periodontology, Center of Dentistry and Oral Medicine, Johann Wolfgang Goethe-University, Frankfurt am Main

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Epping L, Miesbach W, Nickles K, Eickholz P. Is gingival bleeding a symptom of type 2 and 3 von Willebrand disease? PLoS One. 2018 Jan 25;13(1):e0191291. doi: 10.1371/journal.pone.0191291. eCollection 2018. PMID 29370241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the Haemophilia Centre, Medical Clinic III/Institute for Transfusion Medicine, Hospital of the Johann Wolfgang Goethe-University Frankfurt/Main approximately 1500 charts of VWD patients were screened rendering about 35 patients with VWD type 2 and 3.
Pre-assignment Details: From July 16, 2015 to July 15, 2016 24 type 2 and 3 VWD cases were enrolled. Due to the difficulty to find more type 2 and 3 VWD patients willing to participate recruitment was stopped in March 2017 after enrolment of 24 individuals. From April 04, 2016 to March 24, 2017 24 patients that self-reported to be hematologically healthy were enrolled.
Period: Overall Study
Arm/Group | Von Willebrand Disease Type 2 and 3 | Controls
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Von Willebrand Disease Type 2 and 3 | Controls | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (11.8) | 46.6 (12.4) | 46.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of teeth [Mean (Standard Deviation); unit: number of teeth] | 26.7 (2.9) | 26.8 (2.2) | 26.7 (2.5)
current smokers [Number; unit: participants] | 7 | 7 | 14
exhaled carbon monoxide (CO) [Mean (Standard Deviation); unit: ppm] | 3.9 (4.6) | 2.8 (3.4) | 3.4 (4.0)
Pack years (1 pack-year is equal to smoking 20 cigarettes (1 pack) per day for 1 year) [Mean (Standard Deviation); unit: pack years] | 3.3 (6.4) | 1.6 (2.9) | 2.4 (5.0)
Body weight [Mean (Standard Deviation); unit: kg] | 71.6 (16.1) | 68.5 (9.8) | 70.0 (13.3)
HbA1C [Mean (Standard Deviation); unit: percent of gycated hemoglobin] | 5.1 (0.6) | 5 (0.4) | 5.1 (0.5)
Gingivitis [Number; unit: participants] | 11 | 11 | 22
generalized mild, localized moderate chronic periodontitis [Number; unit: participants] | 5 | 5 | 10
generalized mild, localized severe chronic periodontitis [Number; unit: participants] | 3 | 3 | 6
generalized moderate chronic periodontitis [Number; unit: participants] | 2 | 2 | 4
generalized moderate localized severe chronic periodontitis [Number; unit: participants] | 3 | 3 | 6
Von Willebrand antigen [Mean (Standard Deviation); unit: percent] | 44 (45.9) | 122.1 (47.2) | 83.0 (60.6)
Von Willebrand activity [Mean (Standard Deviation); unit: percent] | 24.7 (23.4) | 122.1 (45.1) | 73.4 (60.7)
Factor VIII [Mean (Standard Deviation); unit: percent] | 55.6 (46.3) | 129.8 (27.5) | 92.7 (53.2)
Plaque Control Record [Mean (Standard Deviation); unit: percent] | 53 (24.1) | 49.5 (15.9) | 51.3 (20.3)
activated matrix metalloproteinase 8 (aMMP8) [Number; unit: participants] | 8 | 8 | 16
Probing Pocket Depth [Mean (Standard Deviation); unit: mm] | 1.8 (0.6) | 1.9 (0.5) | 1.9 (0.6)
vertical Probing Attachment Level [Mean (Standard Deviation); unit: mm] | 1.9 (0.7) | 1.8 (1.9) | 1.9 (0.6)
Sum of probing pocket depth (PPD) [Mean (Standard Deviation); unit: mm] | 295 (102.6) | 306.7 (87.6) | 300.8 (94.5)
Sum of PPD with BOP [Mean (Standard Deviation); unit: mm] | 54.4 (37.8) | 49.7 (28.1) | 52.1 (33.0)
Periodontal inflamed surface area [Mean (Standard Deviation); unit: mm²] | 154.4 (124) | 136.1 (95.3) | 145.3 (109.8)
PPD < 4 mm [Mean (Standard Deviation); unit: percent of sites] | 98.5 (3.8) | 98.7 (3.4) | 98.6 (3.6)
PPD 4 to 6.8 mm [Mean (Standard Deviation); unit: percent] | 1.5 (3.8) | 1.3 (3.4) | 1.4 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Bleeding on Probing (BOP)
Description: Using a periodontal probe probing pocket depths (PPD) are assessed with a force of 0.2 N at 6 sites per tooth (mesio-buccal, buccal, disto-buccal, disto-oral, oral, mesio-oral). After 30 seconds bleeding on probing is scored at each site. The frequency of bleeding sites of the total number of assessed sites is calculated as index.
Time Frame: cross-sectional: only one assessment at the time of examination
Measure: Mean (Standard Deviation); unit: percentage of sites
Arm/Group | Von Willebrand Disease Type 2 and 3 | Controls
Number analyzed (Participants) | 24 | 24
percentage of sites | 14.5 (10.1) | 12.3 (5.3)

2. Secondary Outcome: Gingival Bleeding Index (GBI)
Description: A periodontal probe is gently moved through the gingival sulcus. Bleeding is assessed at 6 sites per tooth (mesio-buccal, buccal, disto-buccal, disto-oral, oral, mesio-oral). The frequency of bleeding sites of the total number of assessed sites is calculated as index.
Time Frame: cross-sectional: only one assessment at the time of examination
Measure: Mean (Standard Deviation); unit: percentage of sites
Arm/Group | Von Willebrand Disease Type 2 and 3 | Controls
Number analyzed (Participants) | 24 | 24
percentage of sites | 10.5 (9.9) | 8.8 (4.8)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Von Willebrand Disease Type 2 and 3 | Controls
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
Study is underpowered. A future study may investigate gingival bleeding in VWD and control individuals with more severe periodontal disease. Another interesting question is how hemophilia A and B affect gingival bleeding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT03078595/Prot_SAP_000.pdf